CLINICAL TRIAL: NCT05983250
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Study of Levosimendan in Pulmonary Hypertension Patients With Heart Failure With Preserved Left Ventricular Ejection Fraction (PH-HFpEF)
Brief Title: LEVosimendan to Improve Exercise Limitation in Patients With PH-HFpEF
Acronym: LEVEL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tenax Therapeutics, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-103-06
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Hypertension
Keywords: HFpEF; Pulmonary hypertension group 2; PH-HFpEF; Heart Failure
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blind is maintained by the use of a matching placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- TNX-103 (Active Comparator): oral levosimendan
  Interventions: Drug: TNX-103

INTERVENTIONS:
Drug: TNX-103 — oral levosimendan 1 mg
  Arms: TNX-103
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy of TNX-103 (oral levosimendan) compared with placebo in subjects with PH-HFpEF as measured by the change in 6-Minute Walk Distance (6 MWD; Day 1 to Week 12).

DETAILED DESCRIPTION:
This is a Phase 3, double-blind, randomized, placebo-controlled study of oral levosimendan in patients with PH-HFpEF. There will be a Screening Period of up to 30 days. Subjects will provide written informed consent prior to completing any study procedures. Upon meeting all eligibility criteria, patients will continue to the 12-week randomized, double-blind treatment phase. Approximately 230 subjects will be randomized in a 1:1 ratio to receive an oral dose of levosimendan or placebo

All randomized subjects will have the option to enter the 92-week OLE following the completion of all study events at Week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, greater than or equal to18 to 85 years of age.
2. NYHA Class II or III or NYHA class IV symptoms.
3. A diagnosis of World Health Organization (WHO) Group 2 PH-HFpEF with qualifying hemodynamics
4. Qualifying Baseline RHC.
5. Qualifying echocardiogram
6. Qualifying 6-MWD
7. A 48-hour ambulatory cardiac rhythm monitor during the Screening Period.
8. Requirements related to child bearing potential, contraception, and egg/sperm donation

Exclusion Criteria:

1. A diagnosis of PH WHO Groups 1, 3, 4, or 5.
2. Echocardiographic evidence for hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, cardiac amyloidosis, or infiltrative cardiomyopathy
3. Structural heart repair or replacement of the aortic valve or mitral valve (surgical or percutaneous). OR, planned valve intervention. OR, the presence of significant valve disease
4. A diagnosis of pre-existing lung disease
5. History of severe allergic or anaphylactic reaction or hypersensitivity to the excipients in the investigational product.
6. Major surgery within 60 days.
7. Prior heart, lung, or heart-lung transplants or life expectancy of <12 months
8. History of clinically significant other diseases that may limit or complicate participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in Six-minute walk distance | 12 weeks

SECONDARY OUTCOMES:
KCCQ | 12 weeks
  Change in KCCQ
Clinical Worsening Events | 12 weeks
Change in NT-proBNP | 12 weeks
  Decreases in NT-proBNP may indicate an improvement in symptoms
Change NYHA functional class | 12 weeks
  On a scale of I-IV. Lower scores may indicate improvement in symptoms

CONTACTS AND LOCATIONS:
Locations (40):
- United States (37):
  - Tenax Investigational Site, Tucson, Arizona
  - Tenax Investigational Site, La Jolla, California
  - Tenax Investigational Site, Los Angeles, California
  - Tenax Investigational Site, Sacramento, California
  - Tenax Investigational Site, San Francisco, California
  - Tenax Investigational Site, Torrance, California
  - Tenax Investigational Site, Jacksonville, Florida
  - Tenax Investigational Site, Tampa, Florida
  - Tenax Investigational Site, Winter Haven, Florida
  - Tenax Investigational Site, Atlanta, Georgia
  - Tenax Investigational Site, Chicago, Illinois
  - Tenax Investigational Site, Galesburg, Illinois
  - Tenax Investigational Site, Indianapolis, Indiana
  - Tenax Investigational Site, Louisville, Kentucky
  - Tenax Investigational Site, Boston, Massachusetts
  - Tenax Investigational Site, Minneapolis, Minnesota
  - Tenax Investigational Site, Rochester, Minnesota
  - Tenax Investigational Site, St Louis, Missouri
  - Tenax Investigational Site, Omaha, Nebraska
  - Tenax Investigational Site, New York, New York
  - Tenax Investigational Site, Rochester, New York
  - Tenax Investigational Site, Roslyn, New York
  - Tenax Investigational Site, Charlotte, North Carolina
  - Tenax Investigational Site, Durham, North Carolina
  - Tenax Investigational Site, Greensboro, North Carolina
  - Tenax Investigational Site, Cincinnati, Ohio
  - Tenax Investigational Site, Columbus, Ohio
  - Tenax Investigational Site, Pittsburgh, Pennsylvania
  - Tenax Investigational Site, Providence, Rhode Island
  - Tenax Investigational Site, Charleston, South Carolina
  - Tenax Investigational Site, Columbia, South Carolina
  - Tenax Investigational Site, Dallas, Texas
  - Tenax Investigational Site, Lubbock, Texas
  - Tenax Investigational Site, Plano, Texas
  - Tenax Investigational Site, Murray, Utah
  - Tenax Investigational Site, Richmond, Virginia
  - Tenax Investigational Site, Madison, Wisconsin
- Canada (3):
  - Tenax Investigational Site, Winnipeg, Manitoba
  - Tenax Investigational Site, London, Ontario
  - Tenax Investigational Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No